CLINICAL TRIAL: NCT00950248
Title: Double Blind Placebo-Controlled Phase I/II Clinical Trial of Idebenone in Patients With Primary Progressive Multiple Sclerosis
Brief Title: Clinical Trial of Idebenone in Primary Progressive Multiple Sclerosis (IPPoMS)
Acronym: IPPoMS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 090197; 09-I-0197 (Other: NIH); NCT00950248 (Registry Identifier: clinicaltrials.gov)
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2018-08

CONDITIONS: Primary Progressive Multiple Sclerosis
Keywords: Idebenone; Magnetic Resonance Imaging (MRI); Magnetic Resonance Spectroscopy; Mitochondrial Enhancer; Multiple Sclerosis; MS; Primary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — idebenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- Idebenone (Active Comparator): Idebenone (150mg tablets) administered orally as five tablets, three times per day with food.
  Interventions: Drug: Idebenone
- Placebo (Placebo Comparator): Placebo tablets administered orally as five tablets, three times per day with food.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Idebenone — idebenone, lactose monohydrate, microcrystalline cellulose, croscarmellose sodium povidone, magnesium stearate, silicon dioxide, film-coat: Opadry II 85F23495 (consisting of: aluminium lake, FD&C yellow #6, macrogol/PEG 3550, polyvinylalcohol, titanium dioxide, talc)
  Other Names: SNT-MC17/F02
  Arms: Idebenone
Other: placebo — lactose monohydrate, microcrystalline cellulose, magnesium stearate, film-coat: Opadry II 85F23495 (consisting of: aluminium lake, FD&C yellow #6, macrogol/PEG 3550, polyvinylalcohol, titanium dioxide, talc)
  Other Names: SNT-MC17/F03
  Arms: Placebo

SUMMARY:
Background:

* Multiple sclerosis (MS) is an inflammatory disorder of the central nervous system that progressively weakens and destroys the pathways of the nervous system. About 10 percent to 15 percent of patients develop primary-progressive MS (PP-MS), characterized by progressive accumulation of disability from the disease onset, without any marked improvements or relapses. There are currently no effective treatments for PP-MS.
* Idebenone is a manmade drug that is similar to a naturally occurring compound known as coenzyme Q10, a common dietary supplement. Research data suggest that idebenone may be able to limit demyelination and death of brain cells and thereby slow or halt the progression of neurological dysfunction such as that occurring in MS.

Objectives:

- To evaluate the safety and effectiveness of using idebenone to treat primary progressive MS.

Eligibility:

- Individuals between 18 and 65 years of age who have been diagnosed with primary progressive multiple sclerosis.

Design:

* The study will last 3 years and will be divided into two parts: a 1-year pretreatment baseline and 2 years of treatment with either idebenone or a placebo.
* Pre-treatment study: approximately 5 clinic visits over 1 year.
* Visit 1: Comprehensive medical history and neurological examination, with brain scans and neurological tests.
* Visit 2: Magnetic resonance imaging (MRI) scan of the spine and lymphocytapheresis (withdrawal of white blood cells for testing).
* Visit 3: Lumbar puncture.
* Visit 4: Skin biopsy.
* Visit 5: Repeat MRI of the brain and spinal cord, as well as neurological tests; these tests will be scheduled over 2 days.
* After the five pretreatment visits, patients will receive a 6-month supply of study medication (either idebenone or a placebo) to take three times a day with food
* Patients will continue to have regular followup clinic visits with brain MRI scans, blood tests, and other evaluations of brain and nervous system function. Randomly selected participants will have additional MRI scans for further safety precautions.

DETAILED DESCRIPTION:
Objective: The goal of this study is to assess the safety, therapeutic efficacy and mechanism of action of idebenone in primary-progressive multiple sclerosis (PP-MS) patients.

Study Population: Adult, untreated patients with PP-MS with disability ranging from none to moderately severe will be included in the trial. The upper age limit in this study has been set at 65; setting an age limit should permit us to focus on the potential neuroprotective effect of idebenone in PP-MS and limit the confounding factor of the natural aging process and its known negative influence on neuro-regeneration. Published data indicate that higher doses (10-50 mg/kg) of idebenone per day are required for beneficial effects on neurological disability in comparison to the lower doses (5-10mg/kg) that are sufficient for beneficial effects on cardiac/systemic functions in Friedreich s ataxia (FRDA) patients. Therefore, in order to target the CNS compartment, we will use a daily dose of 2250mg (750mg 3 times per day), which will provide target values of 10-50mg/kg for virtually all adult patients.

Design: This is a Phase I/II safety/efficacy trial with an adaptive trial design: one year of pretreatment baseline period serves the dual purpose of collecting patient-specific biomarkers of disease progression and collecting longitudinal neuroimaging and clinical data for selection of primary outcome measures. This baseline period is then followed by a double-blind, idebenone versus placebo treatment phase for a total of 2 years. Based on preliminary sample size estimates, current enrollment calls for a total of 66 patients (33 per arm).

Outcome Measures: Quantitative neuroimaging measures of central nervous system (CNS: i.e. brain and spinal cord) tissue destruction and clinical and functional (i.e. electrophysiological) measures of neurological disability will be collected every 6-12 months. Additionally, biomarkers focusing on analysis of reactive oxygen species (ROS) and oxidative stress will be collected every 12 months. The trial is currently powered using progression of brain atrophy as detected by SIENA methodology as the primary outcome measure. However, this may not be the most sensitive outcome available. In recognition of this, the trial has an adaptive design: i.e. it incorporates analysis of progression of CNS tissue destruction as measured by quantitative MRI markers and clinical/paraclinical markers defined as secondary outcome measures in the first 30 enrolled patients during the one year pre-treatment baseline, before randomization. All defined outcome measures collected in the first 30 enrolled patients will be transformed into z-scores and compared for the robustness of longitudinal change over the coefficient of variation. This will permit to select the most sensitive and most accurate outcome measure for detecting progression of CNS tissue damage. As a result, the primary outcome measure of this trial will be the comparison of individualized rates of brain atrophy progression between the idebenone and placebo groups after 2 years of treatment, unless the predetermined analysis of the pre-treatment baseline period in the first 30 enrolled subjects determines that one of the predefined secondary outcome measures has a higher z-score than brain atrophy measurement. In this case, the primary outcome would be the efficacy of idebenone versus placebo in inhibiting patient-specific slopes of functional or structural deterioration as measured by this more sensitive biomarker of CNS tissue destruction, yet to be defined by the analysis of the 1-year longitudinal data from pre-treatment baseline.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. PP-MS as determined by the 2005 modification of McDonald s diagnostic criteria
  2. Age from 18-65 years (inclusive)
  3. Expanded Disability Status Scale (EDSS) measure of neurological disability from 1 (no disability, clinical signs only) to 7 (ambulatory with bilateral support)
  4. Able to provide informed consent
  5. Willing to participate in all aspects of trial design and follow-up
  6. If able to become pregnant or to father a child, agreeing to commit to the use of a reliable/accepted method of birth control (i.e. hormonal contraception (birth control pills, injected hormones, vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom with spermicide) or surgical sterilization (hysterectomy, tubal ligation, or vasectomy in a partner)) for the duration of treatment arm of the study
  7. Not receiving any immunomodulatory/immunosuppressive therapies for a period of at least 3 months before enrollment in the study
  8. No exposure to idebenone, coenzyme-Q(10) or other dietary supplements (such as antioxidants, mitochondrial-function promoting supplements or vitamins in excess of 3 times recommended daily doses) for a period of at least 1 month before enrollment in the study

EXCLUSION CRITERIA:

1. Alternative diagnoses that can explain neurological disability and MRI findings
2. Clinically significant medical disorders that, in the judgment of the investigators, could cause CNS tissue damage or limit its repair, or might expose the patient to undue risk of harm or prevent the patient from completing the study
3. History of hypersensitivity reaction to idebenone or coenzyme-Q (10)
4. Pregnant or lactating women. All women of child-bearing potential must have a negative pregnancy test prior to the medication phase of the study.
5. Abnormal screening/baseline blood tests exceeding any of the limits defined below:

   i. Serum alanine transaminase or aspartate transaminase levels greater than 3 times the upper limit of normal values

   ii. Total white blood cell count < 3,000/mm(3)

   iii. Platelet count < 85,000/mm(3)

   iv. Serum creatinine level > 2.0 mg/dl or eGFR (estimated glomerular filtration rate) <30

   v. Positive pregnancy test
6. Patients who are receiving any immunosuppressive therapies (including cytostatic agents) due to the concern that these drugs may contribute to neurodegeneration or limit CNS repair

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bibiana Bielekova, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
raw data will be shared as supplementary material in publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: available at the time of publication

REFERENCES:
- [Background] Artuch R, Aracil A, Mas A, Colome C, Rissech M, Monros E, Pineda M. Friedreich's ataxia: idebenone treatment in early stage patients. Neuropediatrics. 2002 Aug;33(4):190-3. doi: 10.1055/s-2002-34494. PMID 12368988
- [Background] Bielekova B, Catalfamo M, Reichert-Scrivner S, Packer A, Cerna M, Waldmann TA, McFarland H, Henkart PA, Martin R. Regulatory CD56(bright) natural killer cells mediate immunomodulatory effects of IL-2Ralpha-targeted therapy (daclizumab) in multiple sclerosis. Proc Natl Acad Sci U S A. 2006 Apr 11;103(15):5941-6. doi: 10.1073/pnas.0601335103. Epub 2006 Apr 3. PMID 16585503
- [Background] Bieniek M, Altmann DR, Davies GR, Ingle GT, Rashid W, Sastre-Garriga J, Thompson AJ, Miller DH. Cord atrophy separates early primary progressive and relapsing remitting multiple sclerosis. J Neurol Neurosurg Psychiatry. 2006 Sep;77(9):1036-9. doi: 10.1136/jnnp.2006.094748. Epub 2006 Jun 22. PMID 16793860
- [Derived] Kosa P, Ghazali D, Tanigawa M, Barbour C, Cortese I, Kelley W, Snyder B, Ohayon J, Fenton K, Lehky T, Wu T, Greenwood M, Nair G, Bielekova B. Development of a Sensitive Outcome for Economical Drug Screening for Progressive Multiple Sclerosis Treatment. Front Neurol. 2016 Aug 15;7:131. doi: 10.3389/fneur.2016.00131. eCollection 2016. PMID 27574516
- [Derived] Hartung HP, Aktas O. Bleak prospects for primary progressive multiple sclerosis therapy: downs and downs, but a glimmer of hope. Ann Neurol. 2009 Oct;66(4):429-32. doi: 10.1002/ana.21880. No abstract available. PMID 19847907

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 1, 2009 and July 23, 2015, 85 patients were assessed for eligibility and enrolled into the IPPoMS trial at National Institutes of Health, Bethesda, MD
Groups:
- Untreated: Patients in their first year baseline prior to study drug phase
Period: Year 1: Baseline
Arm/Group | Untreated | Idebenone | Placebo
Started | 85 | 0 | 0
Completed | 77 | 0 | 0
Not Completed | 8 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0
Not completed — worsening of symptoms | 2 | 0 | 0
Period: Year 2&3 Treatment Randomization
Arm/Group | Untreated | Idebenone | Placebo
Started | 0 | 39 | 38
Completed | 0 | 33 | 33
Not Completed | 0 | 6 | 5
Not completed — worsening of symptoms | 0 | 2 | 4
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Death | 0 | 0 | 1
Not completed — MRI contraindication | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Idebenone | Placebo | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 37 | 76
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 22 | 18 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 36 | 34 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Age at Disease onset [Mean (Full Range); unit: years] | 43.2 [18.5 to 63.7] | 42.6 [24.2 to 57.5] | 42.9 [18.5 to 63.7]
Time since disease onset at baseline [Mean (Full Range); unit: years] | 13.6 [0.2 to 38.7] | 11.9 [1.6 to 30.1] | 12.7 [0.2 to 38.7]
Body Mass Index [Mean (Full Range); unit: kg/m2] | 25.7 [16.4 to 33.9] | 25.8 [19.9 to 39] | 25.8 [16.4 to 39]
History of Mononucleosis [Count of Participants; unit: Participants]
  Positive | 8 | 6 | 14
  Negative | 19 | 19 | 38
  Unknown | 12 | 13 | 25
Northern European Ancestry [Count of Participants; unit: Participants]
  Positive | 17 | 18 | 35
  Negative | 5 | 5 | 10
  Unknown | 17 | 15 | 32
Family History of MS [Count of Participants; unit: Participants]
  Positive | 13 | 8 | 21
  Negative | 26 | 28 | 54
  Unknown | 0 | 2 | 2
History of Smoking [Count of Participants; unit: Participants]
  Positive | 29 | 30 | 59
  Negative | 9 | 3 | 12
  Unknown | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in the Area Under the Curve (AUC) of the Combinatorial Weight-Adjusted Disability Score (CombiWISE) From Baseline to Treatment Phase
Description: The AUCs of the CombiWISE scores during the 2-year treatment period was analyzed using an Analysis of Covariance (ANCOVA) model with the AUC of the pre-treatment CombiWISE scores, Baseline (Month 0) CombiWISE score and Baseline age as covariates.
  CombiWISE is a composite scale derived from Expanded Disability Status Scale (EDSS) , Scripps Neurological Disability Scale (SNRS), times 25 foot walk (25FW), and non-dominant hand of 9 hole peg test (9HPT) with a minimum value of 0 (no disability) and maximum value of 100 (maximum disability).
  The AUC values were calculated for both the pre-treatment baseline phase (from Months -12, -6, and 0) and for the double-blind phase (from Months 0, 6, 12, 18, and 24).
  Because the follow-up times varied from patient to patient, the AUC values were made comparable by scaling them by dividing the AUC value by the square of the actual duration (in years) of each of the phases.
Time Frame: 1-year pre-treatment baseline vs 2-year treatment period
Population: The primary outcome was assessed in Intention-to-treat population of patients: all randomized patients who have at least one post-baseline (post Mo 0) efficacy assessment. 38 out of 39 patients randomized to idebenone and 35 out of 38 patients randomized to placebo fulfill this definition.
Measure: Mean (Standard Deviation); unit: units on a scale per year
Arm/Group | Idebenone | Placebo
Number analyzed (Participants) | 38 | 35
units on a scale per year | -0.13 (2.17) | -1.04 (2.87)

2. Secondary Outcome: Change in the AUC of Individualized Rates of Enlargement of Ventricular Volume From Baseline to Treatment Phase
Description: The AUCs of the Ventricular volume scores (individualized rates of enlargement of segmented volume of lateral and 3rd ventricles) during the baseline and the 2-year treatment period were assessed using an ANCOVA model with the AUC of the pre-treatment Volumetric score, Baseline (Month 0) Volumetric score, and group as covariates.
  The AUC values were calculated for both the pre-treatment baseline phase (from Months -12, -6, and 0) and for the double-blind phase (from Months 0, 6, 12, 18 and 24).
  Because the follow-up times varied from patient to patient, the AUC values were made comparable by scaling them by dividing the AUC value by the square of the actual duration (in years) of each of the phases.
Time Frame: 1-year pre-treatment baseline vs 2-year treatment period
Population: The primary outcome was assessed in Intention-to-treat population. Due to technical error in MRI images processing 2 out of 38 idebenone patients were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: ml per year
Arm/Group | Idebenone | Placebo
Number analyzed (Participants) | 36 | 35
ml per year | -244 (1094.9) | 35.4382 (1091.1)

3. Secondary Outcome: Disability Progression Measured by EDSS-plus
Description: Categorical time-to-event endpoints (EDSS-plus) were analyzed using Cox Proportional hazards models, with treatment group as a covariate. The EDSS-plus event was defined as disability progression on at least 1 of 3 components [EDSS, 25FW, and/or non-dominant hand 9HPT]) confirmed 6 months apart and with a ≥ 20% minimum threshold change for 25FW and non-dominant hand 9HPT).
  The patients who did not have an event during the study were censored at the time of the last assessment of EDSS-plus. The number of months from the date of first dose to date of event or censoring were used as endpoint. The measure is time to disease progression and unit of this measure is months.
Time Frame: 2-year treatment period
Population: The outcome was assessed in the Intention-to-treat population of patients: all randomized patients who have at least one post-baseline (post Mo 0) efficacy assessment. 38 out of 39 patients randomized to idebenone and 35 out of 38 patients randomized to placebo fulfill this definition.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idebenone | Placebo
Number analyzed (Participants) | 38 | 35
months | 23.1 [12.8 to NA] — the upper limit of the 95% confidence interval cannot be estimated due to insufficient number of participants with events | 23.7 [19.8 to NA] — the upper limit of the 95% confidence interval cannot be estimated due to insufficient number of participants with events

4. Secondary Outcome: Change in Slopes of 25FW Time From Baseline to Treatment Phase
Description: Lower extremity disability was measured by an average of two trials of timed 25 foot walk assessed at month -12, -6, and 0 for the baseline phase and at month 0, 6, 12, 18, and 24 for the treatment phase. The progression rate was calculated as a difference between baseline and treatment slopes using a piecewise linear mixed-effect model with breaking point at month 0.
  The maximum time assigned for a trial is 180s. Patients unable to complete the 25 foot trial within this time limit are coded as "179.9"
Time Frame: 1-year pre-treatment baseline vs 2-year treatment period
Population: The piecewise mixed-effect model only considers patient that completed all follow-up visits, therefore the Completer population (33 patients in placebo and 33 patients in the idebenone group) was considered for this analysis.
Measure: Mean (Standard Error); unit: seconds per year
Arm/Group | Idebenone | Placebo
Number analyzed (Participants) | 33 | 33
seconds per year | 0.02451 (0.01668) | -0.01015 (0.01889)

5. Secondary Outcome: Change in Slopes of 9HPT Time From Baseline to Treatment Phase
Description: Upper extremity/fine motor movements disability was measured as an average of left and right hand time, with each hand assessed as an average of two trials with upper limit of 5 (300s) per trial. Patients unable to complete the task within this time are coded as "777" The outcome was assessed at month -12, -6, and 0 for the baseline phase and at month 0, 6, 12, 18, and 24 for the treatment phase. The progression rate was calculated as a difference between baseline and treatment slopes using a piecewise linear mixed-effect model with breaking point at month 0.
Time Frame: 1-year pre-treatment baseline vs 2-year treatment period
Population: as for outcome 4
Measure: Mean (Standard Error); unit: seconds per year
Arm/Group | Idebenone | Placebo
Number analyzed (Participants) | 33 | 33
seconds per year | 0.001693 (0.000843) | -0.0003 (0.000955)

6. Secondary Outcome: Change in Slopes of SNRS From Baseline to Treatment Phase on
Description: SNRS scale combines various elements of a neurological exam into a single number. The scale ranges from 100 to 0, where 100 marks no disability and 0 marks maximum disability. SNRS was assessed at month -12, -6, and 0 for the baseline phase and at month 0, 6, 12, 18, and 24 for the treatment phase. The progression rate was calculated as a difference between baseline and treatment slopes using a piecewise linear mixed-effect model with breaking point at month 0.
Time Frame: 1-year pre-treatment baseline vs 2-year treatment period
Population: as for outcome 4
Measure: Mean (Standard Error); unit: units on a scale per year
Arm/Group | Idebenone | Placebo
Number analyzed (Participants) | 33 | 33
units on a scale per year | 1.5728 (0.9743) | 0.2315 (0.9702)

7. Secondary Outcome: Change in Slopes of EDSS From Baseline to Treatment Phase
Description: EDSS scale combines various elements of neurological exam. EDSS is a discrete scale ranging from 0 to 10 with 0.5 point increments. EDSS of 0 means no neurological disability, while EDSS of 10 marks death due to MS. EDSS was assessed at month -12, -6, and 0 for the baseline phase and at month 0, 6, 12, 18, and 24 for the treatment phase.The progression rate was calculated as a difference between baseline and treatment slopes using a piecewise linear mixed-effect model with breaking point at month 0.
Time Frame: 1-year pre-treatment baseline vs 2-year treatment period
Population: as for outcome 4
Measure: Mean (Standard Error); unit: units on a scale per year
Arm/Group | Idebenone | Placebo
Number analyzed (Participants) | 33 | 33
units on a scale per year | 1.6148 (3.762) | -3.7879 (3.7214)

ADVERSE EVENTS:
Time Frame: 3 years
Description: First 1 year (Month -12 to Month 0), all patients were untreated - adverse events are reported on all 85 enrolled patients during this pre-treatment phase Next 2 years (Month 0 to Month 24) patients were randomized to placebo (38 patients) or idebenone (39 patients) - adverse events are collected on these 77 patients during the 2 year double-blind phase
Arm/Group | Untreated | Idebenone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/39 | 2/38
Serious Adverse Events (participants affected / at risk) | 12/85 | 11/39 | 10/38
Other Adverse Events (participants affected / at risk) | 28/85 | 15/39 | 11/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Untreated (N=85) | Idebenone (N=39) | Placebo (N=38)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Catheter management (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 1 (1) | 0 (0)
Cholecystectomy (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intrathecal pump insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasticity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Serotonin syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal cord operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia repair (AE) (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Antibiotic therapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Colostomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic hyperglycaemic coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infecti (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Occupational therapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Physical therapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
H1N1 influenza (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Vascular stent occlusion (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Untreated (N=85) | Idebenone (N=39) | Placebo (N=38)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 3 (4) | 3 (4)
Urinary tract infection (Infections and infestations) | 5 (8) | 2 (3) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 3 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Catheter management (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Platelet function test abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increase (Investigations) | 2 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increa (Investigations) | 2 (2) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystectomy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (3) | 1 (1) | 0 (0)
Gravitational oedema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Antiphospholipid antibodies posit (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase abno (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Eye movement disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
General symptom (General disorders) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatic specific antigen increa (Investigations) | 0 (0) | 1 (1) | 0 (0)
Retinal function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Trigeminal nerve ablation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteoperosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase incr (Investigations) | 1 (1) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increas (Investigations) | 1 (1) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ear tube insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Gastritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response sy (General disorders) | 0 (0) | 0 (0) | 1 (1)
Tinea versicolor (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Vasectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Anti-thyroid antibody positive (Investigations) | 1 (2) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increa (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood urine (Investigations) | 1 (1) | 0 (0) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Buttock injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cystoscopy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Glomerular filtration rate increa (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Mean cell volume abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Nuclear magnetic resonance imagin (Investigations) | 1 (1) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Prostate biopsy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The small sample size is a limitation of this study evaluating therapeutic intervention in a complex progressive neurological disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT00950248/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT00950248/SAP_001.pdf